CLINICAL TRIAL: NCT04185454
Title: Estimation of Minimum Efficacy Daily Dose (MTDD) of Jarlsberg Cheese in Healthy Women in Order to Obtain Needed Level of Osteocalcin: A Phase I Dose-finding Study
Brief Title: Estimation of Minimum Efficacy Daily Dose of Jarlsberg Cheese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Stig Larsen (Other)
Collaborators: Tine (Industry)
Responsible Party: Sponsor-Investigator, Prof Stig Larsen, Professor, Meddoc
Organization: Meddoc (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HV-Jarlsberg/IA
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Heathy Women; Pre Menopausal Age; Exlution Criteria: Gastrointestinal Disorder; Liver Disease; Diabetes; Cancer; Kidney Disorder
Keywords: Healthy women; Dose respons; Jarlsberg cheese; Osteocalcin
MeSH Terms: conditions — Liver Diseases; Diabetes Mellitus; Neoplasms; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: The study will be performed as an open, randomised two-dimensional single-centre trial with 3-level between-patient Response Surface Pathway (RSP) design in the first dimension and 3-level within-patient RSP design in the secondary dimension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First design level (Experimental): Three Healthy Voluntary (HV) women were give the same starting daily dose of 100 g Jarlsberg
  Interventions: Dietary Supplement: Jarlsberg cheese
- Second design level (Experimental): Based on the results from the starting dose 5 + 5 HV get a new daily doses of Jarlsberg cheese
  Interventions: Dietary Supplement: Jarlsberg cheese
- Third design level (Experimental): Based on the results from the second design level, the daily dose of Jarlsberg cheese for the next 7 HVs was given
  Interventions: Dietary Supplement: Jarlsberg cheese

INTERVENTIONS:
Dietary Supplement: Jarlsberg cheese — Daily intake of Jarlsberg cheese

SUMMARY:
Aim: To estimate an oral administered recommended minimum efficacy daily dose (MED) of Jarlsberg cheese in order to obtain the needed increased level of Osteocalcin defined as the ratio [Carboxylated / Under Carboxylated] Osteocalcin.

Study population: Healthy Voluntary (HV) women between 20 years and pre-menopausal age.

Design: Open and randomised two-dimensional single-centre trial with 3-level between-patient Response Surface Pathway (RSP) design in the first dimension and 3-level within-patient RSP design in the secondary dimension.

DETAILED DESCRIPTION:
The recruited HV women fulfil the inclusion without the exclusion criteria for the study will undergo a clinical investigation and blood sampling. The participants will be asked to avoid use of other cheese, but eat as usually. One week later, the first clinical investigation will take place including blood sampling. The HV women verified to fulfil the criteria for participation and signed the informed consent form will be included in the study. The trial treatment consisting of a given gr/day Jarlsberg cheese will start the day after this investigation, denoted as Day 0, and the participants receiving a study identification numbers. They will be instructed not to change eating habit except replace use of other chees with Jarlsberg.

The cheese can be consumed with other food at breakfast and/or lunch. The dose of Jarlsberg cheese per day is fixed per participant and varies from 20 gram per day to 180 gram per day with a mid-dose of 100gr/day. The three patients included at the first design level will all receive this mid-dose of 100gr/day. Clinical investigation and blood sampling after start of the treatment, will be performed after 3, 4, and 5 weeks and the ratio [Carboxylated / Under Carboxylated] Osteocalcin will be calculated. This increased Osteocalcin Ratio (OR) based on the results obtained by the blood sampling at week 3 will be classified in five groups and used for determination of the Jarlsberg cheese dose for the five HV women at design level 2. The classifications of increased OR used are: increased OR < 0.5 classifies as Low; 0.5 ≤ increased OR ≤ 0.9 classifies as Moderate Low; 0.9 < increased OR < 1.1 classifies as Suitable; 1.1≤increased OR≤1.5 classifies as Moderate High; increased OR > 1.5 classifies as High. In case the increased OR is found Low or Moderate Low, the daily dose of Jarlsberg cheese will be reduced for the participants at the second design level. If increased OR classifies as Suitable the same dose as at design level 1 will be recommended applied at the second level and if increased OR classifies as moderate High or High, the Jarlsberg cheese-dose will be increased.

The same procedure based on the results obtained from the five participants at the second design level will be used to determine the daily Jarlsberg-dose for the seven HV women at design level 3. With randomization of the recommended cheese-doses at one design level to be used in the next, the between-patient Response-Surface-Pathway (RSP) design-arm is applied.

The within-patient RSP design-arm is applied and related to the duration of the cheese intake. All the participants will consume Jarlsberg cheese during minimum three weeks. Participants obtaining an increased OR ≥ 1 can stop the study. If not, they have to continue until this limit is reached or until maximum five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy voluntary between 20 years and pre-menopausal age

Exclusion Criteria:

* Pregnant women
* Known gastrointestinal disorder
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Lactose intolerance or known milk product allergy
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy voluntary (HV) women
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Osteocalcin ratio | Five weeks
  Ratio between carboxylated and undercarboxylated osteocalcin

SECONDARY OUTCOMES:
Lipid profil 1 | Five weeks
  Triglycerid
Lipid profil 2 | Five weeks
  Cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Helge Lundberg, MD, Principal Investigator — Skjetten Legesenter
Locations (1):
- Skjetten Legesenter, Skjetten, Skedsmo, Norway